CLINICAL TRIAL: NCT04341714
Title: Efficiency and Satisfaction With Telephone Consultation in Neuro-urology: Experience of the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, PHD, Pierre and Marie Curie University
Other Study IDs: GREEN GRC01
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Efficacy, Self; Satisfaction, Patient; Telemedicine
Keywords: telemedicine; neurourology; efficacy; satisfaction
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients enrolled: Patients with telephone consultation on neurourology department, age > 18
  Interventions: Other: Satisfaction evaluation

INTERVENTIONS:
Other: Satisfaction evaluation — Assessement of satisfaction of the telephone consultation

SUMMARY:
The COVID-19 pandemic has necessitated drastic measures in order to limit the spread of SARS-CoV-2. The stay home policies for the whole population and especially for frail patients and the express instruction to deprogram non-urgent consultations and interventions limited the clinic visits in neuro-urology department. In this context, telemedicine was seen as a pragmatic solution to provide follow-up care for our neurologic patients. Due to the delay in deploying telemedicine and the cognitive impairment of some of our patients, telephone consultation has been prioritized.

The COVID-19 pandemic might be an opportunity to review and refine our practices in neuro-urology. For the follow-up of selected patients, telephone consultations may be efficient and cost effective.

The aim of the study is to assess the efficiency and the satisfaction with telephone consultation for the physician and the patient.

The study was conducted in a neuro-urology department of a university hospital in France.

During the stay-home policies for the COVID-19 pandemic, all the scheduled medical visits were converted into telephone consultation. New patients weren't included.

For each teleconsultation, the physician assess the duration of the consultation, the number of tries to join the patient, the efficiency of the consultation, the difficulty to obtain relevant information due to the phone way of the consultation and the lack of physical examination.

On the next days, the patient was contacted by phone and was asked a) if he was satisfied of being phoned by the physician, b) if the teleconsultation was embarrassing, c) if he had enough time of teleconsultation d) if he got all the answers to his queries, e) if he would preferred to had a physical consultation f) to assessed the global satisfaction of the teleconsultation and g) if in the future, they may considered converting some clinic visits to teleconsultations.

The physician and the patient assessed whether this teleconsultation has replaced a physical visit.

The usual transport mode of the patient for a clinic visit and the need to take a day off for worker patients were recorded.

The primary aim was to assess the efficiency and the satisfaction of the telephone consultation. The primary outcome was the evaluation of the efficiency of the telephone consultation by the physician on a numerical 10-points scale. The secondary outcome was the evaluation of the satisfaction of the telephone consultation by the patient on a numerical 10-points scale.

Four hundred teleconsultations are scheduled for five physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Telephone consultation

Exclusion Criteria:

* New patient in the department

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with telephone consultation in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Efficiency of the telephone consultation | 1 day
  The primary outcome was the evaluation of the efficiency of the telephone consultation by the physician on the numeric scale with 0 the worth efficiency and 10 the best efficiency.

SECONDARY OUTCOMES:
Satisfaction of the telephone consultation | 1 day
  The secondary outcome was the evaluation of the satisfaction of the telephone consultation by the patient onon the numeric scale with 0 the worth efficiency and 10 the best efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — Sorbonne Université, GRC 001, GREEN Groupe de Recherche en Neuro-Urologie, AP-HP, Hôpital Tenon, F-75020, Paris, France
Locations (1):
- Department of Neuro- Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided